CLINICAL TRIAL: NCT07332442
Title: Continuous Positive Airway Pressure, Arousability and Links to Mechanisms in Obstructive Sleep Apnea
Acronym: CALM-OSA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); ResMed Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2000040345; 1R01HL179077-01 (NIH)
Record Dates: First submitted 2025-12-23; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Sleep Apnea; Obstructive Sleep Apnea
Keywords: Continuous Positive Airway Pressure (CPAP); sleep apnea; hypnotic; mechanism; arousability
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Eszopiclone

STUDY DESIGN:
Intervention Model Description: randomized, double-blind controlled clinical trial with 3 month follow up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eszopiclone (Experimental): Participants will receive eszopiclone the night of the laboratory split-night polysomnography (PSG, sleep monitoring with and without CPAP therapy). Following polysomnography, participants continue with eszopiclone and CPAP therapy
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator): Participants will receive placebo the night of the laboratory split-night polysomnography (PSG, sleep monitoring with and without CPAP therapy). Following polysomnography, participants continue with placebo and CPAP therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — 3mg for < 65 and 2mg for ≥ 65 years
  Arms: Eszopiclone
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The study design is a randomized, controlled clinical trial to test the hypothesis that arousal threshold (ArTH) will affect how individuals with obstructive sleep apnea (OSA, Apnea-Hypopnea Index (AHI) of 10/hour of higher) respond to CPAP therapy regarding adherence and cognitive function (executive function). Investigators hypothesize that raising ArTH with eszopiclone will improve adherence to CPAP and neurocognitive function with CPAP therapy. Investigators also hypothesize that a lower baseline ArTH is associated with worse CPAP adherence, while a higher baseline ArTH is associated with improved neurocognitive outcomes with CPAP therapy.

DETAILED DESCRIPTION:
Primary Objective The primary objective of this study is to determine whether raising arousal threshold (ArTH) in OSA will improve response to CPAP therapy in people with OSA, where response includes factors such as adherence, change in executive function (Flanker Inhibitory Control test) and cardiovascular function (flow mediated vasodilatation, an exploratory outcome).

Secondary Objective The secondary objective[s] of this study are to understand the mechanisms by which raising ArTH may improve adherence to CPAP, neurocognitive and cardiovascular function. The mechanisms investigated include sleep duration, depth, CPAP level and tolerance, hypoxia, patient symptoms, biomarkers of neuronal damage, oxidative stress and sympathetic activation.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Clinically confirmed new diagnosis of OSA:

  1. Polysomnography AHI ≥ 10 per hour of sleep and/or
  2. Home sleep apnea testing, respiratory even index, REI ≥ 10 per hour of recording

Exclusion Criteria:

* Known non-OSA related conditions associated with sleep-disordered breathing (e.g., a central disorder of hypersomnolence, neurological, neuromuscular, or pulmonary disorder)
* Use of sleep-inducing medications (e.g., other non-benzodiazepine sedative hypnotic-drugs [e.g., zoldpidem], benzodiazepines, non-selective antihistamines, trazodone, opiates, barbituates)
* Known hypersensitivity reaction to eszopiclone
* Contraindications to its use based on medical history or function (e.g., dizziness at baseline or established mobility problems or imbalance)
* History of complex sleep behaviors (e.g., NREM or REM parasomnias)
* Concomitant use of ≥ 2 servings of alcohol per night or other CNS depressant for 2 weeks prior or throughout the study
* Sleep opportunity of less than 7 hours
* Severe active depression or other mental health disorders (e.g., schizophrenia, bipolar disorder, personality disorder).
* History of sleep-walking, sleep-driving, and engaging in other activities while not fully awake
* Severe hepatic impairment (liver function tests 2 X the upper limit of normal)
* Unstable medical condition (e.g., decompensated heart failure, end-stage chronic obstructive pulmonary disease, end-stage renal disease)
* Females of childbearing potential who are pregnant, breastfeeding, or intend to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
CPAP adherence | Daily over 3 months
  Mean daily average of CPAP use over 3 months
Flanker inhibitory control and attention test | Baseline, 1-, 2- and 3-months
  Executive function is assessed using the validated NIH Toolbox Cognition Battery's Flanker inhibitory control and attention test. In a Flanker task, participants are required to indicate the left-right orientation of a centrally presented stimulus while inhibiting attention to the potentially incongruent stimuli that surround it (i.e., the flankers, typically two on either side). Primary outcome is the overall percent of correct responses in incongruent trials.

SECONDARY OUTCOMES:
Mean Epworth Sleepiness Scale score Scores | Baseline, 1-, 2-and 3-months
  Sleep questionnaire of subjective sleepiness. Total score range of 0-24; scores above 10 suggest excessive sleepiness.
Mean Functional Outcomes of Sleep Questionnaire (FOSQ) short form score | Baseline, 1-, 2-and 3-months
  Measures how sleepiness affects daily life, with scores ranging from 5-20. Higher scores indicate better functioning and less impairment.
Mean Insomnia Severity Index score (ISI) Scores | Baseline, 1-, 2-and 3-months
  ISI is a validated 7-question survey. The total score range is 0-28 with higher scores indicating more severe insomnia.
Mean PROMIS Sleep Disturbance score Scores | Baseline, 1-, 2-and 3-months
  T-score mean of 50 and a standard deviation (SD) of 10. Higher scores indicating more sleep disturbance.
Mean PROMIS Sleep-Related Impairment score Scores | Baseline, 1-, 2-and 3-months
  T-score mean of 50 and a standard deviation (SD) of 10. Higher scores indicating more sleep disturbance.
Mean time to complete Trail Making Test (TMT) A and B | Baseline, 1-, 2-and 3-months
  Administered on standardized paper form by research associate. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper and participant connect numbers (Part A) and numbers with letters (Part B) in ascending order. Mean time to connect the "trail" in minutes.
Mean processing speed of Pattern Comparison Processing Speed Test | Baseline, 1-, 2-and 3-months
  Administered by participants via an iPad to assess processing speed. Participants are asked to quickly determine whether two stimuli are the same or not the same. Mean time in seconds.
Mean reaction time of Psychomotor vigilance test (PVT) | Baseline, 1-, 2-and 3-months
  Administered by participants via a computer to complete psychomotor vigilance task at the same time in the morning. Mean time in minutes to complete assessment of daytime vigilance = 1/reaction-time.
Mean percent accuracy of Change Card Sort Test | Baseline, 1-, 2-and 3-months
  Administered by participants via an iPad to assess cognitive flexibility and attention. The participant is asked to match a series of picture pairs to a target picture.
Mean percent correct recall of Verbal Paired Associates A-B task | Baseline and 3-months
  Administered by participants via an iPad with audio instructions and feedback to assess recall. The participant is asked to recall A-B verbal paired associates word-pairs. Immediate recall occurs before sleep and delayed recall occurs after sleep.
Mean OSA alleviation at 3 months | 3 months
  Defined as: therapeutic efficacy × adjusted CPAP adherence. The therapeutic efficacy for OSA is "[AHI-baseline - AveAHI-3-months on CPAP] / AHI-baseline" and the adjusted CPAP adherence is objective AveCPAP use / AveSleep time (both in hours) over 3 months
Mean percent hypoxic burden | Baseline and at the night of CPAP and eszopiclone/placebo initiation: 3 weeks after baseline visit
  Hypoxic burden (HB) is a sleep apnea metric that quantifies the total oxygen deprivation by measuring the depth and duration of blood oxygen drops (desaturations) during sleep, expressed as %-minutes per hour.
Mean sleep depth score | Baseline and at the night of CPAP and eszopiclone/placebo initiation: 3 weeks after baseline visit
  Sleep depth will be measured by an Odds Ratio Product (ORP), a continuous metric based on quantitative analysis of the EEG power spectra. High values indicate deeper sleep, with a range of 0 - 2.5.
Arousal intensity | Baseline and at the night of CPAP and eszopiclone/placebo initiation: 3 weeks after baseline visit
  Arousal intensity is measured on a scale between 0 and 9 (most intense) using a validated automated wavelet transformation method (Azarbarizin et al., Sleep 2014)
Ventilatory burden | Baseline and at the night of CPAP and eszopiclone/placebo initiation: 3 weeks after baseline visit
  The average ventilatory burden per event is defined as the multiplication of the average ventilation during the respiratory event (i.e., event depth) and average duration of respiratory events. The total ventilatory burden (percentage eupnea × min/h) for each participant is defined as the multiplication of respiratory event rate (events/h) and average ventilatory area per event (percentage eupnea × min/event).
Mean concentration Neurofilament Light Chain (NfL) | Baseline and 3-months
  Mean concentration NfL (pg/ml) in the blood to assess neuronal injury and damage.
Mean concentration Aβ40 | Baseline and 3-months
  Mean concentration Aβ40 (pg/ml) in the blood (usually measured as a ratio with Aβ42 (Aβ42/40 ratio) to assess brain amyloid plaque buildup.
Mean concentration F2-isprostane | Baseline and 3-months
  Mean concentration F2-isprostane (pg/ml) in the blood to assess oxidative stress.
Mean concentration oxidized LDL | Baseline and 3-months
  Mean concentration oxidized LDL (pg/ml) in the blood to assess oxidative stress.
Mean morning concentration cortisol | Baseline and 3-months
  Mean concentration cortisol (pg/ml) in the blood to assess autonomic activation.
Mean concentration norepinephrine | Baseline and 3-months
  Mean concentration norepinephrine (pg/ml) in the blood to assess autonomic activation.
Mean systolic and diastolic blood pressure (BP) | Baseline and 3-months
  Mean systolic and diastolic blood pressure during a single 24-hour period at baseline and 3-month
Blood pressure variability | Baseline and 3-months
  Blood pressure variability during a single 24-hour period at baseline and 3-month
Mean nighttime BP dipping | Baseline and 3-months
  Mean nighttime BP dipping during a single 24-hour period at baseline and 3-month
Mean CPAP pressure over 3 months | Assessed daily over 3 months
  Measured nightly from cloud-based remote monitoring adherence system
Mean residual AHI over 3 months | Assessed daily over 3 months
  Measured nightly from cloud-based remote monitoring adherence system

OTHER OUTCOMES:
Flow mediated vasodilation (FMD) - exploratory | baseline and 3 months
  FMD is a standard non-invasive technique for assessing endothelial function. FMD will be obtained using a standard method by a trained RA at the same time of the day after the baseline PSG and the 3-month follow-up. Two-dimensional longitudinal images will be acquired using Doppler ultrasound to assess arterial diameter and flow velocity (resting and hyperemic). Resting blood flow is estimated by time-averaging the pulsed Doppler signal obtained from a mid-vessel sample volume. The blood pressure cuff is then inflated to >50 mmHg above systolic pressure to occlude arterial inflow for 5 minutes. A cuff is then deflated, and a pulse wave and longitudinal images are obtained at 10 seconds and 60 seconds (hyperemia). The FMD is the percent increase in vessel diameter from baseline to hyperemia.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Zinchuk,, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale Centers for Sleep Medicine, North Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No